CLINICAL TRIAL: NCT07062614
Title: Exploration of Intra-individual Variability of Exposure to Emtricitabine and Lamivudine in Hair With a View to Validating the Value of This Matrix as a Diagnostic Tool for Partial and/or Total Non-compliance With Antiretroviral Treatment
Brief Title: Exploration of the Variability of Exposure to Antiretroviral Treatment in Hair With a View to Validating Its Value as a Diagnostic Tool for Partial and/or Total Non-compliance With Treatment
Acronym: HAIROBS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0574; ID-RCB (Other: 2025-A00212-47)
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: Antiretroviral treatment; hair; intra-individual variance; HIV; Human immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lamivudine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Lamivudine treatment: HIV patients who are on treatment with Lamivudine
  Interventions: Other: Hair sampling and questionnaires answers for Patients with Lamivudine or Emtricitabine treatment
- Patients with Emtricitabine treatment: HIV patients who are on treatment with Emtricitabine
  Interventions: Other: Hair sampling and questionnaires answers for Patients with Lamivudine or Emtricitabine treatment

INTERVENTIONS:
Other: Hair sampling and questionnaires answers for Patients with Lamivudine or Emtricitabine treatment — at inclusion, 3 months and 6 months of follow-up, patients must answer the Girerd compliance questionnaire. After 6 months of follow-up, two strands of hair will be taken from the base of the skull using scissors

SUMMARY:
Treatment adherence is defined by compliance with the dosage schedule (i.e., dose per dose and number of doses per day), as well as the duration of administration (i.e., number of days during which the dosage schedule must be followed).

Treatment adherence determines the therapeutic efficacy and the absence of toxicity of the prescribed medication. However, this adherence is far from being respected even by patients with serious pathologies such as patients living with HIV (PLWHIV). However, among PLWHIV, non-adherence is a significant source of virological failure and is difficult to assess because it is most often based on what the patient reports to their doctor. A currently used approach consists of determining the drug concentration in the blood and possibly that of its metabolite(s). However, determining a drug's blood concentration presents two major pitfalls: (i) it is necessary to take a blood sample, which remains an invasive procedure for the patient; (ii) for the vast majority of drugs, if the patient scrupulously adheres to the dosage schedule a few days before the blood sample is taken, the drug concentration is most often within the expected range. Therefore, a concentration in the reference range does not exclude partial or even total non-compliance between two medical visits. Saliva is a more easily accessible matrix than blood. However, the same representativeness problem is encountered due to the fact that saliva is in almost instantaneous equilibrium with blood.

Urine could be used to assess compliance. However, this requires multiple urine collections between two doses. This constraint is not compatible with the organization of clinical services. The objective is to determine intra-individual variability in the amount of antiretroviral (ARV) in different segments of the same strand of hair during periods of full treatment adherence.

This objective is preliminary to the use of hair as a tool for detecting treatment non-adherence in patients.

Two reference antiretroviral molecules will be documented: Emtricitabine and Lamivudine, as they are present, one or the other, in the majority of antiretroviral combination strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient living with HIV
* Patient receiving stable antiretroviral therapy (i.e., no change in treatment strategy or dosage regimen) for at least 6 months.
* Patient receiving antiretroviral therapy based on emtricitabine or lamivudine.
* Patient identified as compliant based on patient follow-up data: (i) patient's reported adherence to the infectious disease physician (i.e., simple self-report), (ii) virological data (i.e., absence of blips in the last 18 months), (iii) pharmacological data (i.e., plasma antiretroviral concentrations within the expected range) if concentrations were previously measured as part of the patient's follow-up.
* Patient agreeing not to cut their hair to less than 6 cm of remaining length during the 6 months of the study.
* Patient agreeing to have their hair sampled at the end of the 6 months.
* Patients over 18 and under 70 years of age.
* Individuals who have not objected.
* Individuals enrolled in the French Health Insurance

Exclusion Criteria:

* Pregnant women.
* Patients planning to color/bleach their hair in the next 6 months.
* Patients planning to have their hair straightened/restyled in the next 6 months.
* Persons under judicial protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HIV and receiving antiretroviral therapy with Emtricitabine or Lamivudine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Individuality index for each patient | 6 months after the inclusion
  Determine the individuality index for each patient, defined as:
  ID = 1 - (intra-individual variance) / (inter-individual variance) with intra-individual variance being the variation in ARV concentrations in different segments of the same strand of hair within a patient, and inter-individual variance being the variation in ARV concentrations in hair between patients. An individuality index less than 0.2 means that the variability within an individual is as great as that found in a population of individuals treated with the same antiretroviral, i.e., the distribution of this antiretroviral in the hair is too variable to make hair a good tool for assessing adherence.

SECONDARY OUTCOMES:
Ratio of the mean hair concentration to the plasma antiretroviral concentration | 6 months after the inclusion
  Ratio, for each included patient, of the mean hair concentration (over 6 months) to the plasma antiretroviral concentration determined at the 6-month hair collection visit.
Mathematical model describing the relationship between blood and hair | 6 months after the inclusion
  Nonlinear mixed-effect mathematical/statistical model describing the relationship between blood and hair
Rate of refusal to participate in the study | 6 months after the inclusion
  Number of people who refused to participate in the study because of hair sampling to estimate the difficulties of implementation in a hospital setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious and Tropical Diseases Department, Purpan University Hospital, Toulouse Place du Docteur Baylac, Toulouse, France

IPD SHARING:
Plan to Share IPD: No